CLINICAL TRIAL: NCT04226274
Title: A Phase 1b, Open-label Study to Evaluate the Safety and Tolerability of 12 Weeks Treatment With Oral REN001 in Patients With McArdle Disease (Glycogen Storage Disorder 5)
Brief Title: A Study of the Safety of REN001 in Patients With McArdle Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reneo Pharma Ltd (Industry)
Responsible Party: Sponsor
Organization: OnKure, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REN001-103
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: McArdle Disease
MeSH Terms: conditions — Glycogen Storage Disease Type V

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REN001 (Experimental): Oral
  Interventions: Drug: REN001

INTERVENTIONS:
Drug: REN001 — Once daily for 12 weeks

SUMMARY:
The purpose of this study is to assess REN001 safety in subjects with McArdle Disease

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give written, signed and dated informed consent
* Confirmed diagnosis of McArdle Disease
* Subjects must be able to remain on stable medication through the study and specifically must not commence or have changes to agents that affect metabolism such as medication for diabetes
* Follow a stable dietary regimen as documented by a 3-day dietary record obtained during the screening period.

Exclusion Criteria:

* Documented history of ongoing rhabdomyolysis
* Evidence of acute crisis from their underlying disease
* Currently following or planning to start a ketogenic diet
* Treatment with an investigational drug within 1 month or within 5 half-lives, whichever is longer
* Have been hospitalized within the 3 months prior to screening for any major medical condition
* Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator in discussion with the Medical Monitor, would make the subject inappropriate for entry into this study
* Pregnant or nursing females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
Adverse Events | up to Week 12
  Number of participants with Adverse Events (AEs) as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Rosaline Quinlivan, MD, Principal Investigator — MRC Centre for Neuromuscular Diseases, London
Locations (2):
- Instituto de Investigación Hospital 12 de Octubre, Madrid, Spain
- National Hospital for Neurology and Neurosurgery, Queens Square, London, United Kingdom